CLINICAL TRIAL: NCT00695682
Title: The Safety and Tolerability of Intravitreal Infliximab (Remicade) in Patients With Refractory Diabetic Macular Edema or Choroidal Neovascularization Secondary to Age Related Macular Degeneration- A Pilot Study
Brief Title: Intravitreal Infliximab for Diabetic Macular Edema (DME) and Choroidal Neovascularization (CNV)
Acronym: ITVR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Retina Research Foundation (Other)
Responsible Party: Paul Beer, MD, Retina Research Foundation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101606
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Diabetic Retinopathy; Macular Degeneration
Keywords: Remicade; Infliximab; CSME; BDR; CNV; AMD
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intravitreal injection of infliximab — All subjects will receive 0.5 mg/ 0.05 mL of infliximab by intravitreal injection at their first treatment visit or the 6 weeks visit if eligible for a repeat injection.

SUMMARY:
Injections of medicine into the middle of the eye (intravitreal injections) are commonly used in a multitude of retinal diseases. We are looking for new treatments that may be beneficial in treating retinal disease and improving patients' vision.

Infliximab (Remicade) is a genetically engineered antibody against a molecule in the body called TNF-α. It neutralizes the effects of TNF-α by binding to it. Intravenous Infliximab has been used for inflammatory arthritic conditions and Crohn's disease since 1998. We do not know if infliximab injections into the eye are safe. We are performing this pilot study to determine if they can be safe.

DETAILED DESCRIPTION:
Intravenous Infliximab is currently used for the treatment of systemic inflammatory conditions and inflammatory disease of the eye with a relatively favorable safety profile. However, systemic administration carries the risk of systemic side effects, which in the case of infliximab can be severe, such as increased risk of infection, reactivation of tuberculosis or Hepatosplenic T-cell Lymphoma.

Direct intravitreal administration of medication is the preferred method of treatment for retinal vascular disorders. The eye is a self contained organ relatively isolated from the systemic circulation by the tight blood retinal barrier. Effective intraocular drug levels can be achieved with a much smaller amount of medication if injected intravitreally and this also results in minimal systemic exposure to the patient. Preliminary studies have shown that Infliximab may have a positive role in the management of retinal vascular disorders in humans when administered intravenously, and can be an effective treatment intravitreally in animal models. No data has been published yet on intravitreal use of infliximab in human subjects.

We plan to study the safety and tolerability of intravitreal injections of infliximab in human subjects with refractory diabetic macular edema or choroidal neovascularization. Our infliximab dose will be 0.5mg/0.5ml, as it follows the reconstitution instructions in the Product Insert. This dosing will fall within the therapeutic dosing found within the animal study as it leads to the same vitreous concentration as the7.5 µg dose in group B rat eye study. (4)

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 21 years
* Patients with active CNV secondary to AMD in the study eye which did not improve with conventional therapy
* Patients with refractory diabetic macular edema in the study eye which did not improve with conventional therapy
* BCVA 20/70 or less as measured on an ETDRS chart.

Exclusion Criteria:

* Are participating in another clinical study requiring follow up examinations
* Have received any other experimental drug within 12 weeks prior to enrollment
* Are unwilling or unable to follow or comply with all study-related procedures
* Inability to obtain photographs, fluorescein angiography, or optical coherence tomography to document CNV, e.g. due to media opacity, allergy to fluorescein dye or lack of venous access
* Aphakia or pseudophakia with the absence of posterior capsule (unless it resulted from a yttrium aluminum garner [YAG]) posterior capsulotomy)
* Within two months prior to screening, have had intraocular surgery (including cataract surgery) in the study eye
* Within 1 month prior to screening had YAG laser in the study eye
* Have had intravitreal anti VEGF or intravitreal steroids in the last 6 weeks
* Have had previous pars plana vitrectomy in the study eye
* Are pregnant or are trying to become pregnant
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Have a history of allergies to murine monoclonal antibodies, mice or mouse products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
This is a pilot study to study the safety and tolerability of intravitreal Infliximab in patients with refractory diabetic macular edema and choroidal neovascularization (CNV) | 3 m

SECONDARY OUTCOMES:
(BCVA) | 3m
Standard Electroretinogram | 3m
OCT | 3m
Fluorescein angiography | 3m
Nidek Microperimetry | 3m
Incidence and severity of adverse events | 3m

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Beer, MD, Principal Investigator — Retina Research Foundation
Locations (1):
- Retina Consultants, Slingerlands, New York, United States

REFERENCES:
- See also: Retina Research Foundation — http://retinaresearchfoundation.org
- See also: Retina Consultants — http://retinaconsultants.org